CLINICAL TRIAL: NCT04552977
Title: A Trail of Fluzoparil in Combination With Temozolomide in Patients With Recurrent Glioblastoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, President of Shandong Cancer Hospital and Institute, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GBM-IIT-SHR3162-TMZ
Record Dates: First submitted 2020-09-14; First posted 2020-09-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Glioblastoma
Keywords: glioblastoma, fluzoparil
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fluzoparil+temozolomide (Experimental): Participants receive fluzoparil and temozolomide
  Interventions: Drug: fluzoparil; Drug: temozolomide

INTERVENTIONS:
Drug: fluzoparil — a PARP1 inhibitor
Drug: temozolomide — an alkylating chemotherapeutic agent

SUMMARY:
This is a one arm, open, single center phase II study. The main purpose of this study was to evaluate the efficacy and safety of fluzoparil combined with temozolomide in patients with recurrent glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and written informed consent;
2. The age was 18-70 years old, with no gender limit;
3. Supratentorial space occupying lesions were diagnosed as glioblastoma by pathology;
4. Patients received standard radiotherapy and temozolomide concurrent chemotherapy after surgery, and the interval between the last radiotherapy and the last radiotherapy was ≥ 4 weeks (pseudo progression should be excluded);
5. MRI confirmed that the tumor had definite recurrence. The diameter of the enhancement focus was more than 1 cm and more than 2 layers (layer spacing was 5 mm), or the recurrence was confirmed by pathology after re biopsy or operation;
6. The recurrence site or other reasons can not be resected;
7. The methylation status of MGMT promoter had been detected or was willing to be detected before enrollment;
8. According to recist1.1, there was at least one measurable lesion;
9. KPS score ≥ 60 points;
10. The tablets can be swallowed normally;
11. The expected survival time was more than 3 months;
12. Sufficient organs and bone marrow function. The definition is as follows.

    1. Neutrophil count (ANC) ≥ 1500 / mm3 (1.5 ×109 / L);
    2. Platelet count (PLT) ≥ 100000 / mm3 (100 × 109 / L);
    3. Hemoglobin (HB) ≥ 9 g / dl (90 g / L);
    4. Serum albumin ≥ 2.8 g / dl;
    5. Serum creatinine ≤ 1.5 times the upper limit of normal value (ULN) or creatinine clearance rate ≥ 60 ml / min;
    6. Total bilirubin (TB) ≤ 1.5 × ULN, or total bilirubin (TB) > 1.5 × ULN, but direct bilirubin (DBIL) ≤ 1 × ULN; patients with liver metastasis should be ≤ 2 × ULN;
    7. The level of AST / SGOT or ALT / SGPT should be ≤ 2.5 × ULN and ≤ 5 × ULN in patients with liver metastasis;
    8. Left ventricular ejection fraction (LVEF) ≥ 50%, QTc < 450 ms in male and < 470ms in female;
13. The international normalized ratio (INR) of prothrombin time was ≤1.5 and activated partial thromboplastin time (APTT) were ≤1.5 times the upper limit of normal value in patients who had not received anticoagulant therapy. Patients receiving full dose or parenteral anticoagulant therapy can enter the clinical trial as long as the dosage of anticoagulant drugs is stable for at least 2 weeks before entering the clinical study, and the results of coagulation test are within the limits of local treatment;
14. Women of childbearing age should have negative pregnancy test (serum or urine) within 7 days before enrollment, and voluntarily use appropriate contraceptive methods during the observation period and within 8 weeks after the last administration of the study drug; for men, it should be surgical sterilization or agree to use appropriate contraceptive methods during the observation period and within 8 weeks after the last administration of the study drug;
15. Good compliance, can cooperate with the study and follow-up according to the requirements of the program.

Exclusion Criteria:

1. Patients had been treated with PARP inhibitors in the past;
2. Previous allergic history of temozolomide or fluzoparide, previous allergy to dacarbazine, and allergic reaction to temozolomide or fluzoparide;
3. Patients had inherited galactose intolerance, lactase deficiency and glucose galactose malabsorption;
4. The following treatments or drugs were received before the first study treatment:

   1. Major surgery (biopsy is allowed due to diagnosis) or severe trauma within 4 weeks before the first use of the study drug;
   2. Received strong CYP3A4 inducer or inhibitor within 2 weeks after the first use of the study drug;
   3. Previously vaccinated with anti-tumor vaccine; vaccinated with live attenuated vaccine within 28 days before the first study drug treatment or within 60 days after the end of study drug treatment;
5. Currently participating in other clinical studies, unless it is an observational (non intervention) clinical study or an intervention in the follow-up of a new clinical study; or has participated in any other drug clinical study within 4 weeks before the first administration, or no more than 5 half-life from the last study medication;
6. Except basal cell carcinoma or squamous cell carcinoma of skin, superficial bladder cancer, carcinoma in situ of cervix, intraductal carcinoma in situ of breast and papillary thyroid carcinoma which can be treated locally and have been cured in the past 5 years or at the same time;
7. Advanced patients with symptoms, spread to the viscera, and at risk of life-threatening complications in a short period of time (including patients with uncontrollable large amount of exudate [chest, pericardium, abdominal cavity];
8. Fever of unknown origin > 38.5℃ occurred during the screening period / before the first administration (according to the researcher's judgment, fever caused by tumor can be included in the group);
9. Severe infection (CTCAE > Level 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infection complications, etc. the baseline chest imaging examination revealed active pulmonary inflammation, symptoms and signs of infection within 2 weeks before the first use of the study drug, or the need for oral or intravenous antibiotic treatment (excluding prophylactic use of antibiotics)；
10. Within 6 months before entering the study, the following conditions occurred: myocardial infarction, severe / unstable angina pectoris, NYHA grade 2 or above cardiac insufficiency and clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention; hypertension with poor drug control (systolic blood pressure continuously increased ≥ 150mmhg or diastolic blood pressure ≥ 100mmhg);
11. History of gastrointestinal bleeding or tendency of gastrointestinal bleeding in the past 6 months, such as esophageal varices, local active ulcer lesions, fecal occult blood≥(+) (gastroscopy is required when fecal occult blood is (+));
12. Unable to swallow the study drug, chronic diarrhea (including but not limited to irritable bowel syndrome, Crohn's disease, ulcerative colitis), intestinal obstruction and other factors affecting drug administration and absorption;
13. Urine protein ≥ + + + or 24-hour urine protein > 1.0g;
14. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation or congenital immunodeficiency was known;
15. Patients with active pulmonary tuberculosis infection found through medical history or CT examination, or patients with active pulmonary tuberculosis infection within one year before enrollment, or patients with active pulmonary tuberculosis infection history one year ago but without regular treatment;
16. Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS); untreated active hepatitis B (hepatitis B, defined as hepatitis B virus surface antigen [HBsAg] positive test results, HBV-DNA ≥ 500 Hepatitis C was defined as hepatitis C antibody [HCV AB] positive, HCV-RNA higher than the detection limit of analysis method and abnormal liver function), or combined with hepatitis B and hepatitis C co infection;
17. Patients had a clear history of neurological or mental disorders, including epilepsy and dementia, and was known to have a history of psychotropic substance abuse, alcoholism or drug abuse;
18. Patients who were considered unsuitable for the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
6-months PFS rate in all participants by RECIST 1.1 | Up to approximately 24 months
  6-months progression-free survival rate in all participants by RECIST 1.1

SECONDARY OUTCOMES:
ORR in all paients by RECIST Version 1.1 | Up to approximately 24 months
  ORR was assessed by performing study imaging every 6-9 weeks after the first dose of study treatment. ORR was defined as the proportion of participants in the analysis population who had a CR defined as a disappearance of all target lesions with pathological lymph nodes having a reduction in short axis to <10 mm) or PR defined as at least a 30% decrease in the sum of diameters of target lesions, using the baseline sum diameters as a reference.
Disease control rate in all patients by RECIST Version 1.1 | Up to approximately 24 months
  Disease control rate is defined as the proportion of patients whose best curative effect reaches complete remission, partial remission or disease control. Maintain for at least 4 weeks by RECIST Version 1.1
Overall survival (OS) in all participants | Up to approximately 24 months
  OS was defined as the time from the first day of study treatment to death due to any cause. OS was analyzed by the Kaplan-Meier method for censored data and reported in months.
mPFS in all participants | Up to approximately 24 months
  mPFS was defined as as the median time from the first day of study treatment to the first documented PD per RECIST 1.1 or death due to any cause, whichever occurred first.
mOS in all participants | Up to approximately 24 months
  mOS was defined as the time from the first day of study treatment to death due to any cause.
Number of participants experiencing an adverse event (AE) | From first dose to last dose of treatment plus 2 months of follow-up, up to 24 months
  An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product/protocol-specified procedure, whether or not considered related to the medicinal product/protocol-specified procedure. Any worsening of a preexisting condition temporally associated with the use of the product was also an AE. A serious adverse event (SAE) was an AE that resulted in death, was life threatening, resulted in persistent or significant disability/incapacity, resulted in or prolonged an existing inpatient hospitalization, was a congenital anomaly/birth defect, was a cancer, was associated with an overdose, was another important medical event.
Number of participants experiencing a serious adverse event (SAE) | From first dose to last dose of treatment plus 2 months of follow-up, up to 24 months
  Any event which causes death, permanent damage, birth defects, or requires hospitalization is considered an SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, Ph.D, M.D, Principal Investigator — Shandong Cancer Hospital and Institute

IPD SHARING:
Plan to Share IPD: No